CLINICAL TRIAL: NCT05604378
Title: Does Epstein-Barr Virus-positive Gastric Cancer Establish a Significant Relationship With the Multiple Genes Related to Gastric Carcinogenesis?
Brief Title: Relationship of EBV-positive Gastric Cancer and Multiple Genes Associated With Gastric Carcinogenesis
Status: Completed | Type: Observational
Sponsor: Saint Vincent's Hospital, Korea (Other)
Responsible Party: Sponsor
Other Study IDs: VC22RISI0177
Record Dates: First submitted 2022-10-28; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-08

CONDITIONS: Gastric Cancer; EBV Infection; MSI
Keywords: Gastric Cancer; EBV; MSI; Prognosis
MeSH Terms: conditions — Stomach Neoplasms; Epstein-Barr Virus Infections | interventions — Gastrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EBV-positive gastric cancers
  Interventions: Procedure: Gastrectomy
- EBV-negative gastric cancers
  Interventions: Procedure: Gastrectomy

INTERVENTIONS:
Procedure: Gastrectomy — All patients in our study underwent gastrectomy.

SUMMARY:
The data of 460 gastric cancer patients who underwent curative gastrectomy with D2 lymph node dissection between January 2017 and February 2022 were analyzed. The clinicopathological features and prognosis of the patients with EBV-positive gastric cancers were compared with those of EBV-negative gastric cancers. Immunohistochemistry for epidermal growth factor receptor (EGFR), C-erb B2, Ki-67, and p53 was performed. Additionally, in situ hybridization was conducted to detect EBV, and microsatellite instability (MSI) analysis was used to assess the deficiency in mismatch repair (MMR) genes.

DETAILED DESCRIPTION:
This study collected consecutively the data of 463 patients with gastric adenocarcinomas who underwent curative gastrectomy with lymphadenectomy at our institution between January 2017 and February 2022. The Institutional Review Board of St. Vincent's Hospital, The Catholic University of Korea approved this study (VC22RISI0177). Informed consent of the patients was waived because of the retrospective nature of the study. The inclusion criteria were: (1) gastric adenocarcinoma; (2) R0 resection; (3) formalin-fixed paraffin-embedded tissue (FFPE) blocks available for analysis. Patients who had undergone previous surgery, palliative resection, chemotherapy, or radiation therapy were excluded. All patients underwent gastrectomy with lymphadenectomy based on the Korean Practice Guideline for Gastric Cancer 2018 [18]. After the surgery, clinical follow-up data were collected every 6 months during the first year and then every year thereafter. Disease-free survival (DFS) was defined as the length of time from curative surgery to the first tumor recurrence or distant metastasis. Overall survival (OS) was defined as the time from curative surgery to death from any cause.

ELIGIBILITY:
Inclusion Criteria:

* (1) gastric adenocarcinoma; (2) R0 resection; (3) formalin-fixed paraffin-embedded tissue (FFPE) blocks available for analysis.

Exclusion Criteria:

* Patients who had undergone previous surgery, palliative resection, chemotherapy, or radiation therapy were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study collected consecutively the data of 463 patients with gastric adenocarcinomas who underwent curative gastrectomy with lymphadenectomy at our institution between January 2017 and February 2022.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
EBV positive gastric cancer is associated with increased Ki-67 and decreased EGFR. | Between January 2017 and February 2022.

CONTACTS AND LOCATIONS:
Overall Officials: Kyong Hwa Jun, Ph.D., Study Director — The Catholic University of Korea
Locations (1):
- Jiwon Seo, Suwon, Gyeong-Gi-Do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided